CLINICAL TRIAL: NCT01794442
Title: Correlation Between Retinal Metabolism and the Observation of a Visible Retinal Spontaneous Venous Pulse
Brief Title: Study on the Oxygen Saturation in Pulsating and Non-pulsating Central Retinal Veins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S120213
Record Dates: First submitted 2013-02-12; First posted 2013-02-18 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2013-01

CONDITIONS: Open Angle Glaucoma; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controls: Healthy volunteers with no family history of glaucoma, an increased or asymmetrical cup/disc ratio or any other optic disc structural change (notching, disc hemorrhage) or an intraocular pressure (IOP) above 21 mmHg that could suggest possible glaucoma suspects.
- Primary open-angle glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at least one measurement of IOP of >21 mmHg required
- Normal Tension Glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at maximum recorded IOP of < 21 mmHg

SUMMARY:
Retinal ischemia is thought to play an important role in the pathogenesis of glaucoma. Recent findings have confirmed that there is a direct correlation between the levels of venous oxygen saturation and the degree of the glaucomatous disease, presumably due to a decrease in retinal cell metabolism.

However, glaucoma patients have been suggested to have a different pattern in retinal venous circulation. For instance, the observation of a visible pulsating central retinal vein is a phenomenon that can be seen in up to 98% of the healthy individuals but is identifiable in less than 50% of glaucoma patients. While the nature of these venous changes are not year clear, the lack of a visible pulsating flow could suggest an increased intraluminal venous pressure due to some obstruction from both ocular or extraocular structures. This undetermined increase in venous pulse pressure could then significantly decrease perfusion pressures and therefore further decrease oxygen supply to the retinal tissues.

The investigators will therefore try to determine if there is a significant difference between the oxygen saturation of the retinal vessels in both glaucoma patients with and without a visible pulsating central vein

DETAILED DESCRIPTION:
1. Visual field examen will be performed.
2. Structural examination of the optic disc (confocal microscopy) will be performed.
3. Spontaneous venous pulsation will be recorded after a one minute fundoscopy observation.
4. Oximetry reading in the non-contact retinal oximetry of the first 3 order retinal vessels

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years old
* willing to sign an informed consent and able to comply with the requirements of the study
* having no other ocular diseases besides glaucoma

Exclusion Criteria:

* history of ocular trauma
* intraocular surgery (except for cataract surgery)
* eye disease (except glaucoma)
* systemic diseases with ocular involvement like diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Retinal Oxygen saturation in retinal veins with absent pulsation | Up to 3 months
  We will assess, through analysing the oximetry recordings from both pulsating and non-pulsating retinal veins, whether there are any differences in venous or arterial-venous oxygen saturation in primary open-angle glaucoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, ND, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium